CLINICAL TRIAL: NCT07011121
Title: Determine the Clinical Effectiveness of Mobile CenteringPregnancy to Improve Maternal and Infant Health Outcomes of Marshallese in Arkansas
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2P20GM109096-06 (NIH); 2P20GM109096-06 (NIH)
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Prenatal Care
Keywords: Marshallese; CenteringPregnancy

STUDY DESIGN:
Intervention Model Description: . Using a Hybrid Type 1 effectiveness-implementation trial; the proposed study will establish approaches to determine the preliminary effectiveness of an innovative, culturally adapted, Mobile CenteringPregnancy program to improve prenatal care attendance and the early-stage impact on improved knowledge, attitudes, and behaviors. Additionally, we will establish approaches to determine the effectiveness of Mobile CenteringPregnnacy to improve preterm birth (primary outcome) and maternal outcomes (secondary outcomes): low-birth weight and breastfeeding initiation for Marshallese women. We will also assess implementation outcomes and identify key implementation determinants, which will inform the design of strategies to support wider implementation of the program. A Hybrid Type 1 is the correct study design because we do not yet have robust data on the effectiveness of delivery Mobile CenteringPregnancy to Marshallese women, and both implementation outcomes and determinants are unknown. O
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group prenatal care (Experimental): . CenteringPregnancy, a group prenatal care model, is a promising alternative that challenges the standard model of one-on-one prenatal counseling. Previous research has documented that group prenatal care is associated with a lower prevalence of preterm birth and low birth weight infants. 18,39 Group prenatal care also has been associated with improved maternal mental health, breastfeeding, optimal pregnancy weight gain, improved postpartum weight loss, better birth spacing, and higher patient satisfaction. 18,39 All participants will attend routine one-on-one prenatal appointments prior to the intervention. The sessions occur from week 14 of pregnancy through birth with women of similar gestational age, following the same schedule as standard care. Once the groups of women are formed (5 per group), the participants attend all appointments together for the duration of their pregnancies. Mobile health clinic located at FBOs will provide a location for providers to provide brief one-on
  Interventions: Behavioral: CenteringPregnancy

INTERVENTIONS:
Behavioral: CenteringPregnancy — . CenteringPregnancy, a group prenatal care model, is a promising alternative that challenges the standard model of one-on-one prenatal counseling. Previous research has documented that group prenatal care is associated with a lower prevalence of preterm birth and low birth weight infants. 18,39 Group prenatal care also has been associated with improved maternal mental health, breastfeeding, optimal pregnancy weight gain, improved postpartum weight loss, better birth spacing, and higher patient satisfaction. 18,39 All participants will attend routine one-on-one prenatal appointments prior to the intervention. The sessions occur from week 14 of pregnancy through birth with women of similar gestational age, following the same schedule as standard care. Once the groups of women are formed (5 per group), the participants attend all appointments together for the duration of their pregnancies. Mobile health clinic located at FBOs will provide a location for providers to provide brief one-on-

SUMMARY:
Pacific Islanders bear a disproportionate burden of obesity compared to other racial/ethnic minorities and the United States (US) population. Pacific Islanders residing in the US also have high maternal and infant health disparities with disproportionally high rates of preterm birth (<37 weeks) and low birthweight infants (<2,500 grams). They are also more likely to experience preeclampsia, primary cesarean birth, excessive gestational weight gain, gestational diabetes mellitus, and low exclusive breastfeeding rates compared to other racial/ethnic minorities and the US population in general. These unique health circumstances increase medical complications and are associated with impaired glucose intolerance, delivery complications, and higher incidence of obesity and metabolic disease risk later in life for infants. Early and consistent supportive care throughout the pregnancy continuum is strongly associated with positive birth outcomes that can mitigate childhood obesity.

However, Pacific Islanders are less likely to receive adequate prenatal care compared to other racial and/or ethnic minorities. Our preliminary studies using Arkansas birth records (n=2,488; 2019) have shown that Marshallese experience exceptionally poor perinatal outcomes, even compared to other US Pacific Islanders. Specifically, 15% of Marshallese women received no prenatal care (compared to 1.6% women nationally); more than 50% do not attend the recommended number of prenatal care visits; 19% of Marshallese infants were born preterm (compared to 9.6% nationally); and 15% of Marshallese infants were low birthweight (compared to 8.3% nationally). These poor health outcomes are highly associated with childhood obesity risk through increased odds of rapid infant weight gain and sub-optimal infant feeding practices. Thus, our foundational work demonstrates an urgent need for culturally adapted interventions to engage the Marshallese community in Arkansas in prenatal care that optimize birth outcomes that can mitigate childhood obesity.

CenteringPregnancy, an evidenced-based group prenatal care model, challenges the standard model of one- on-one prenatal counseling and has demonstrated effectiveness in other populations in lowering the risk of preterm birth, low birthweight infants, and increasing exclusive breastfeeding initiation compared to women receiving individualized care. Our prior work has demonstrated how challenging delivering group care is to the Marshallese community because of transportation barriers. Mobile health clinics are transforming the US healthcare system by delivering services directly to communities of need. However, mobile health clinics have not yet been implemented with group prenatal programs like CenteringPregnancy in the US. The proposed study will determine the preliminary effectiveness of an innovative Mobile CenteringPregnancy program for Marshallese women while also evaluating implementation determinants and outcomes to inform sustainable scaling of the program.

DETAILED DESCRIPTION:
Overview. Using a Hybrid Type 1 effectiveness-implementation trial; the proposed study will establish approaches to determine the preliminary effectiveness of an innovative, culturally adapted, Mobile CenteringPregnancy program to improve prenatal care attendance and the early-stage impact on improved knowledge, attitudes, and behaviors. Additionally, the investigators will establish approaches to determine the effectiveness of Mobile CenteringPregnnacy to improve preterm birth (primary outcome) and maternal outcomes (secondary outcomes): low-birth weight and breastfeeding initiation for Marshallese women. Investigators will also assess implementation outcomes and identify key implementation determinants, which will inform the design of strategies to support wider implementation of the program. A Hybrid Type 1 is the correct study design because the investigators do not yet have robust data on the effectiveness of delivery Mobile CenteringPregnancy to Marshallese women, and both implementation outcomes and determinants are unknown. Our chosen approach also balances scientific rigor and community needs. Investigators will use an external control approach with a propensity score matched comparison group. Investigators considered a two-arm randomized controlled trial, but our community advisors did not feel it was ethical given the stark needs.

In Aim 1, investigators will use a mixed-methods approach to examine adherence to prenatal care appointments and the early-stage impact on knowledge, attitudes, and behaviors at pre-intervention and post-intervention. In Aim 2, investigators will establish key statistical approaches to determine the effectiveness of Mobile CenteringPregnancy to improve preterm birth (primary outcome) and maternal health outcomes (secondary outcome) that promote healthy development and mitigate childhood obesity in infants. A birth certificate data review will be used to document preterm birth, low-birth weight infants, and breastfeeding initiation in the intervention arm and the matched control group. In Aim 3, investigators will assess implementation outcomes and multilevel determinants of implementation and sustainability of Mobile CenteringPregnancy. Using a mixed methods design, investigators will assess implementation of the intervention using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) evaluation framework. This study will demonstrate the preliminary effectiveness of a culturally adapted Mobile CenteringPregnancy intervention. Further, these aims are in direct response to reviewer comments from a scored NIH RO1 on Mobile CenteringPregnnacy. The data collected from this proposed study will provide the necessary preliminary results to design a larger trail.

ELIGIBILITY:
Inclusion Criteria:

* (1) women who self-report as Marshallese
* (2) 18 years of age or older
* (3) pregnant (12-14 weeks gestation; confirmed with ultrasound).

Exclusion Criteria:

* (1) conception with the use of fertility treatments
* (2) high-risk pregnancy that requires a transfer to a high-risk clinic
* (3) multiple gestations (i.e. pregnant with more than one infant)
* (4) use of medications known to influence fetal growth (e.g., glucocorticoids, insulin, thyroid, hormones).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
pre-term birth | three months postpartum
  birth prior to 36 weeks gestation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Community Health Innovation, Springdale, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
All data will be aggregated when disseminated to provide confidentiality to all participants.